CLINICAL TRIAL: NCT05619965
Title: Awake Endotracheal Intubation With Glidescope Video Assisted Laryngoscope vs Fiberoptic Bronchoscope in Patients With Traumatic Cervical Injury; Randomized Controlled Trial
Brief Title: Awake Endotracheal Intubation in Cervical Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mona Mohamed Mogahed, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 35636/8/22
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Trauma; Patient Satisfaction; Airway Morbidity
MeSH Terms: conditions — Wounds and Injuries; Patient Satisfaction | interventions — Hypnotics and Sedatives

STUDY DESIGN:
Intervention Model Description: The investigators will compare awake endotracheal intubation with glidescope video assisted laryngoscope vs fiberoptic bronchoscope in patients with traumatic cervical injury
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Awake Glidoscope Videolaryngoscope (Active Comparator): Awake endotracheal intubation of cervical trauma patients by Glidoscope Videolaryngoscope
  Interventions: Drug: sedative; Device: Awake endotracheal intubation by Glidescope videolaryngoscope
- Awake Fiberoptic bronchoscope (Active Comparator): Awake endotracheal intubation of cervical trauma patients by Fiberoptic bronchoscope
  Interventions: Drug: sedative; Device: Awake endotracheal intubation by Fiberoptic bronchoscope

INTERVENTIONS:
Drug: sedative — dexmedetomidine 1 mic/kg IV over 10 minutes then 0.4 mic/kg/h continuous IV infusion
Device: Awake endotracheal intubation by Glidescope videolaryngoscope — Awake endotracheal intubation by Glidescope videolaryngoscope of cervical trauma patient
  Arms: Awake Glidoscope Videolaryngoscope
Device: Awake endotracheal intubation by Fiberoptic bronchoscope — Awake endotracheal intubation by Fiberoptic bronchoscope of cervical trauma patient
  Arms: Awake Fiberoptic bronchoscope

SUMMARY:
The researcher will compare awake endotracheal intubation with glidescope video assisted laryngoscope vs fiberoptic bronchoscope in patients with traumatic cervical injury;

DETAILED DESCRIPTION:
One hundred patients undergoing post traumatic cervical spine fixation under general anesthesia will be randomly allocated to two groups in a prospective study. Between December 2022 and May 2023.

All patients will be premedicated before the procedure and after giving 500 ml of lactated ringer solution with glycopyrrolate 0.2 mg iv and dexmedetomidine 1 mic/kg IV over 10 minutes then 0.4 mic/kg/h continuous IV infusion. All patients will receive standard clinical care monitoring including three lead ECG, noninvasive arterial blood pressure measurement and pulse oximeter. Patient will be administered oxygen 6 L/min through nasal prong.

Patients will be allocated into two equal groups (50 patients per group) for awake intubation with either FOB (F group) or GVL (G group) according to computer generated randomization technique. Each patient will receive nebulization with 5 ml of lidocaine 1% for 5 min followed by topicalization of soft palate and fauces with 5 puffs of lidocaine spray (10 mg/spray) immediately before the technique of endotracheal intubation (ID 6.5 mm for female and 7 mm in male, armored tube. Before airway manipulation each patient will receive a bolus dose of fentanil 1 mic/kg.

During the procedure Philadelphia cervical collar will be removed and MILS of cervical spine will be carried out by trained assistant (senior registrar anesthetist, 5 years' experience). After successful intubation (by consultant anesthesia who had more than 100 times successful intubation with either FOB or GVL) and neurological assessment (by spinal surgeon), general anesthesia will be induced with propofol 1.5 mg/kg, cisatracurium 0.1 mg/kg and remifentanil 0.5 lg/kg. Hypotension (decreased in MAPP 20% of base line) will be treated with ephedrine bolus 5-10 mg and 250 ml of lactated ringer solution. Only three attempts will be permitted per each patient and if failed plan B was to carry out endotracheal intubation under inhalational induction with FOB without neuromuscular blockade and to exclude patients from the study. Attempt will be held if O2 saturation decreased below 90%.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients
* ages 26-44
* undergoing a selective cervical spine fixation.

Exclusion Criteria:

* body mass index (BMI) more than 35 kg/m2.
* Obstructive airway disease
* cardiovascular disease
* apparent airway difficulty
* patient refusal .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
intubating time | immediately post endotracheal intubation
  (defined as the time from introduction of the scope till confirmation of correct endotracheal tube placement with three waves endtidal capnography)
intubating attempts | immediately post endotracheal intubation
  intubating attempts per each patient (will be recorded by dedicated technician).

SECONDARY OUTCOMES:
heart rate | immediately post endotracheal intubation
mean arterial blood pressure | immediately post endotracheal intubation
patient satisfaction (score; excellent =1, good =2 and fair = 3). | immediately post endotracheal intubation
  (score; excellent =1, good =2 and fair = 3).